CLINICAL TRIAL: NCT00346372
Title: Optical Coherence Tomography of Retinal Abnormalities Associated With Choroidal Nevus, Choroidal Melanoma and Choroidal Melanoma Treated With Iodine-125 Brachytherapy
Status: Terminated | Type: Observational
Why Stopped: low accrual
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: UCLA IRB#03-11-052
Record Dates: First submitted 2006-06-27; First posted 2006-06-29 (Estimated); Last update posted 2019-08-12 (Actual); Status verified 2018-01

CONDITIONS: Ocular Melanoma
Keywords: Ocular Melanoma; Optical Coherence Tomography; Eye Tumor; Choroidal Melanoma; Uveal Melanoma
MeSH Terms: conditions — Uveal Melanoma; Eye Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
During regularly scheduled appointments, Optical Coherence Tomography (OCT) is performed on consented subjects. The OCT is a new type of camera that takes very detailed pictures inside of the eye and deeper into eye tissues. Optical Coherence Tomography imaging of intraocular tumors may lead to improved diagnosis and monitoring of tumors within the eye.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years or older) with:

  * choroidal nevus greater than or equal to 3.0 mm in longest basal diameter, or greater than or equal to 1.25 mm in apical height or:
  * choroidal melanoma located in the posterior pole (4mm or less from the center of fovea or the border of the optic nerve head)

Exclusion Criteria:

* Ocular media opacity in the tumor eye that prevents adequate functional testing or imaging and prior or concurrent retinal or choroidal disease in the tumor eye that prevents adequate functional testing or imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who meet the following Eligibility Criteria
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2004-03; Primary Completion 2017-11-27 (Actual); Study Completion 2017-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley R Straatsma, MD, JD, Principal Investigator — Jules Stein Eye Institute, UCLA
Locations (1):
- Jules Stein Eye Institute, Los Angeles, California, United States